CLINICAL TRIAL: NCT04324229
Title: Liraglutide in the Prevention of Type 2 Diabetes After Gestational Diabetes
Acronym: Liragest
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Heidi Immonen, Principal Investigator, Consultant in Endocrinology, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T160/2018
Record Dates: First submitted 2020-03-15; First posted 2020-03-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- liraglutide (Active Comparator)
  Interventions: Drug: Liraglutide 6 MG/ML [Victoza]
- placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Liraglutide 6 MG/ML [Victoza] — Starting dose of liraglutide 0.6 mg will be administered for one week, after which dose will be escalated to liraglutide 1.2 mg for one week and thereafter liraglutide 1.8 mg s.c. daily injections.
  Arms: liraglutide
Drug: Placebos — Starting dose of placebo 0.1 ml will be administered for one week, after which dose will be escalated to placebo 0.2 ml for one week and thereafter placebo 0.3 ml s.c. daily injections.
  Arms: placebo

SUMMARY:
Obese women with history of gestational diabetes are in great danger to develop type 2 diabetes (T2D) within 5-10 years after delivery. Aim of the study is to investigate if 12 months' liraglutide treatment could decrease the risk of T2D in obese women who have had gestational diabetes. The women are randomized either to liraglutide (Victoza ® 1.8 mg) or placebo group, once daily. Same laboratory tests are taken and instructions given at baseline 6 month and one year. After one year visits once a year until 5 years with same laboratory tests and measurements are taken.

DETAILED DESCRIPTION:
Incidence of type 2 diabetes (T2D) is increasing along with pandemia of obesity. Gestational diabetes is the major risk factor for T2D in women and more than every tenth will develop gestational diabetes during pregnancy. T2D can be prevented by weight loss. Health care professionals should take advantage of this opportunity to prevent this devastating disease in women.

Aim of the study is to investigate if 12 months' liraglutide treatment (1.8 mg) once daily could decrease the risk of T2D in obese women who have had gestational diabetes needing treatment with metformin and/or insulin.

100 women, who have had gestational diabetes with treatment with metformin and/or insulin and who have stopped lactation and are not pregnant are enrolled between 6 to 18 months after delivery. BMI should be ≥30 kg/m2. The women are randomized either to liraglutide (Victoza ® 1.8 mg) or placebo group. Both treatments are given by similar device s.c. once daily during 365 days. Before starting the treatment, clinical examination and laboratory test are done. Similar dietary instructions are given. Same laboratory tests are taken and instructions given at 6 months and at one year after baseline. Additional follow-up call (AE reporting) is scheduled at 3 months and a drug dispensing visit at 9 months. After one year visits once a year until 5 years with same laboratory tests and measurements are taken. Primary end-point is development of T2D (fasting P-glucose >7 mmol/l and/ or 2 h >11 mmol/l in oral glucose tolerance test 75g, and/or HbA1c≥ 6.5 %) from year 1 to 5.

ELIGIBILITY:
Inclusion Criteria:

* history of gestational diabetes with treatment with metformin and/or insulin
* delivery 6 to 18 months before screening
* BMI ≥30 kg/m2
* use of contraceptives (IU-device or oral contraceptive)

Exclusion Criteria:

* lactation
* pregnancy
* type 1 or type 2 diabetes
* use of antidepressives, statins or anti-hyperglycemic therapies
* severe hepatic insufficiency
* end stage renal disease
* history of pancreatitis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes | from year 1 to 5
  assessed by fasting P-glucose >7 mmol/l and/ or 2 h >11 mmol/l in oral glucose tolerance test (OGTT) 75g, and/or HbA1c≥ 6.5 %

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided